CLINICAL TRIAL: NCT06379841
Title: Comparing Operative Times in Hysteroscopies With Full Draping vs Green Draping
Brief Title: Green Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael Heit, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00007357
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hysteroscopy
Keywords: Surgical Draping; Hysteroscopy Draping; Draping Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Draping (Experimental): This arm will follow the green draping procedures.
  Interventions: Procedure: Green Draping Procedure
- Full Draping (Active Comparator): This arm will follow the conventional full draping procedures.
  Interventions: Procedure: Full Draping Procedure

INTERVENTIONS:
Procedure: Green Draping Procedure — The green draping will include only an under-buttock. After normal hand hygiene and scrub, the green draping procedure will have the surgeons don only a single pair of sterile gloves.
  Arms: Green Draping
Procedure: Full Draping Procedure — The full draping will include under-buttocks, two-leg drapes, blue towels, and a top drape. After normal hand hygiene and scrub, the draping procedure will have the surgeon don a surgical gown and two sets of sterile gloves for the surgeon.
  Arms: Full Draping

SUMMARY:
The purpose of this study is to determine whether green draping in the operating room prior to a hysteroscopy results in a decreased operating room time.

Secondary aims are to determine whether there are any differences in infection rate, complication rate, fluid deficit, operating room turnover time

DETAILED DESCRIPTION:
Climate change will affect global health, with a disproportionate effect on women. To continue advocating for the patient population, it is necessary to decrease the carbon footprint of the medical field. The healthcare industry is responsible for many carbon emissions and waste generation. In a hospital, the operating room contributes 20-30% and uses 3-6 times more energy per square foot. There are growing attempts at "green" strategies to minimize the carbon footprint of surgery. Parts of this strategy include decreasing the amount of single-use supplies. From its production, transport, use, and disposal life cycle, single-use supplies contribute to a large amount to waste.

Hysteroscopies are a very common procedure with over 200,00 performed per year. hysteroscopy involves placing a camera into the uterus via the vagina and cervix. This can be performed for both diagnostic and therapeutic indications. Hysteroscopies have been classically performed in the operating room. In the operating room, there is an emphasis on maintaining the sterile field. The patient is prepped and draped, resulting in a large amount of excess drape usage. However, in-office hysteroscopies are gaining in popularity. In the office, draping is limited to the under buttock to capture the efflux. Institutions such as Newton Wellesley Hospital and Medstar Hospital systems all utilize minimal draping in the in-office setting.

There is no further sterile draping. There is not an increased risk of infections from in-office hysteroscopies. Overall, the rate of infections from hysteroscopy is very low ranging from 0.06- 0.18%. A study has shown that the usage of preoperative iodine in hysteroscopic in-office procedures does not decrease the postoperative infection rate. New studies focused on a minimal drape cystoscopy have also not shown any increase in infection rate.

The investigator and the team hypothesize that green draping for a hysteroscopy can decrease the operative time of a procedure without causing increased complications. This will also add to the procedure's decreased cost and carbon footprint.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing a hysteroscopic procedure at Emory St Joseph's, Emory Dunwoody ASC, Emory University Hospital, Emory University Hospital ASC.

Exclusion Criteria:

* Women undergoing a concomitant procedure along with the hysteroscopic procedure
* Pregnant women,
* Prisoners
* Cognitively impaired or Individuals with impaired decision-making capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Difference in operative times | Baseline
  The principal investigator will begin timing the case on a stopwatch when the surgeon has finished scrubbing and reentered the operating room. The investigator will note the end time of the procedure as when the procedure has concluded, and the patient's legs are brought out of lithotomy back onto the bed.

SECONDARY OUTCOMES:
Infection Rate | Baseline, 2 weeks
  De-identified case report forms will be used for collection of perioperative data including total Infection rate.
Post Operative complication Rate | Baseline, 2 weeks
  De-identified case report forms will be used for collection of Post operative data including urinary tract infection, vaginal infection, intrauterine infection, abnormal postoperative bleeding.
Peri operative Complication Rate | Baseline, 2 weeks
  De-identified case report forms will be used for collection of perioperative data including total complication rate. The complication rate is a composite to include uterine perforation, fluid overload, hemorrhage, and air/gas embolism.
Number of cases of Fluid deficits | Baseline, 2 weeks
  De-identified case report forms will be used for collection of data including total number of patients with fluid deficits.
Operative room turnover time in Full Draping | Baseline
  The OR turnover time will be calculated from the operating room status board as the difference between when the patient is out of the room and when the next patient is brought into the room.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Heit, MD,PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Hospital, Atlanta, Georgia
  - Emory Dunwoody Clinic, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT06379841/ICF_000.pdf